CLINICAL TRIAL: NCT06349083
Title: Neurobehavioral Mechanisms of Psilocybin-assisted Treatment for Alcohol Use Disorder
Brief Title: Neurobehavioral Mechanisms of Psilocybin-assisted Treatment for AUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-01227; 5R01AA031417-02 (NIH)
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: psilocybin; AUD
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral high-dose of psilocybin (Experimental): Participants will receive a single IP administration session of psilocybin (30 mg total) and three supportive therapy sessions.
  Interventions: Drug: Psilocybin; Behavioral: Supportive therapy sessions
- Placebo control (Placebo Comparator): Participants will receive a single IP administration session of matching placebo capsules and three supportive therapy sessions.
  Interventions: Other: Inactive Placebo; Behavioral: Supportive therapy sessions

INTERVENTIONS:
Drug: Psilocybin — One 25 mg capsule and one 5 mg capsule (30 mg total) administered once orally
  Arms: Oral high-dose of psilocybin
Other: Inactive Placebo — Two matching placebo capsules administered once orally
  Arms: Placebo control
Behavioral: Supportive therapy sessions — Participants will receive three supportive therapy sessions of manual-based treatment from a Center for Psychedelic Medicine (CPM) clinician, accompanied by a Silver Hill Hospital (SHH) therapist who has an ongoing therapeutic relationship with the participant. The CPM clinician will be a licensed physician, clinical psychologist, or nurse practitioner who will be solely responsible for the content of the intervention. The SHH therapist will provide additional support and continuity with clinical treatment.

SUMMARY:
This is a double-blind, randomized, placebo-controlled Phase 2 mechanistic clinical trial designed to evaluate the therapeutic neural mechanisms of psilocybin in patients with alcohol use disorder (AUD), and to determine whether further studies are warranted to study the relationship of any such effects to clinical improvement in AUD symptoms. The primary aims are to evaluate the effects of psilocybin on AUD; measures will include 1) fMRI neural activation and functional connectivity, using a well-validated task to characterize neural and subjective response to negative affective and alcohol visual stimuli; 2) alcohol use data (self-report and blood biomarkers); and 3) self-report measures related the NE, IS, and EF domains.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide voluntary informed consent
2. Have a breath alcohol concentration (BrAC) ≤ 0.01% at screening, as determined by a breath alcohol reading from a calibrated breath alcohol sensor. (Note: this criterion may be re-evaluated within the 30-day screening period. This criterion will also be reassessed at Baseline, on Day 0, and on Day 2. Those not meeting the criterion may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator).
3. Are able to read, speak, and understand English, as documented during the informed consent process.

   a. Non-English speaking subjects will be excluded because the study is using only validated English-language versions of assessment instruments.
4. Are 18 to 65 years old, inclusive, at Screening visit.
5. Have DSM-5 diagnosis of moderate or severe Alcohol Use Disorder (AUD) (using MINI)
6. Are in treatment at Silver Hill Hospital (either in Residential Treatment program, or Inpatient with plan to enter Residential Treatment Program)
7. Are able and willing to adhere to all study requirements, including attending all study visits and therapy sessions, and completing all assessments.
8. Have least 4 heavy drinking days (4 or more drinks per day for a woman, 5 or more drinks per day for a man) in the 30 days prior to admission to SHH
9. Agree to refrain from any non-prescribed psychotropic substance or illicit drug use for at least 72 hours prior to investigational product (IP) administration, and for at least 24 hours before each fMRI assessment visit, with the exceptions of nicotine and caffeine. Regarding nicotine, they must agree not to use nicotine for at least 1 hour before and 6 hours following IP administration, and for at least 1 hour before fMRI scans. Regarding caffeine, they must agree to consume approximately their usual amount of caffeine on the morning of Day 0 (prior to IP administration).
10. Agree to refrain from taking all non-prescription medications and supplements (nutritional and herbal) for at least 1 week prior to the IP administration session unless approved by the Investigator.
11. Are able to swallow capsules.
12. Have a negative pregnancy test at screening, Baseline, Day 0 (pre-IP administration); and Day 2.
13. If able to become pregnant or produce viable sperm (male or female), are willing to use approved contraception for duration of the trial
14. Able to provide at least 2 locators.

Exclusion Criteria:

1. Pregnancy or lactation
2. Any medical condition that would preclude safe participation in the study, including the following, as determined by medical history review, physical examination, electrocardiogram (ECG), and clinical laboratory tests:

   a. Seizure disorder ii. Significantly impaired liver function, defined as 1) alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); 2) ALT or AST > 3 × ULN with concomitant total bilirubin > 2.0 × ULN; or 3) ALT or AST ≥ 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia.

   iii. Cardiovascular disease including coronary artery disease, angina, history of arrhythmia (unless a successful ablation has been performed), heart failure, history of heart valve replacement, and history of cerebrovascular accident or transient ischemic attack.

   iv. Uncontrolled hypertension with systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg. (Note: participants who otherwise qualify at the Screening visit will have 3 opportunities to produce 1 blood pressure reading ≤ 140/90 mmHg (each reading will be collected at least 15 minutes apart). If blood pressure the Screening visit is consistently elevated > 140/90 mmHg across all 3 attempts, participants may be referred to their primary care provider for management of hypertension. Upon management of blood pressure, participants will have an opportunity to return once within the 30 day screening window to make 3 additional attempts at a blood pressure reading ≤ 140/90 mmHg. Participants will be considered eligible upon registering 1 blood pressure reading ≤ 140/90 mmHg during the Screening period.) v. Resting heart rate > 100 bpm (Note: participants will have an opportunity to return once within the 30 day screening window to make 3 additional attempts at a resting heart rate ≤ 100 bpm.).

   vi. Serious ECG abnormalities present on the ECG obtained on Day -65 (e.g., evidence of ischemia, myocardial infarction, QT interval corrected for heart rate [QTc] prolongation (QTc > 0.450 seconds), arrhythmia, or conduction abnormalities that increase the risk of arrhythmia.

   vii. Hyperthyroidism viii. Insulin-dependent diabetes ix. Any other medical condition which precludes safe participation in the study in the medical opinion of the Investigator. (Note: medical history will be updated on Day 0. Those not meeting the criterion will not be randomized but may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
3. Have any of the following DSM-5 psychiatric disorders, as determined by the MINI and Psychiatric History AT the Screening Visit: (Note: psychiatric history will be re-evaluated on Day 0, but the MINI will not be re-administered on Day 0)

   1. Lifetime history of schizophrenia spectrum or other psychotic disorder (including substance or medication-induced psychosis or psychosis due to a co-occurring medical condition).
   2. Current alcohol withdrawal (CIWA-Ar score >7)
   3. History of mania
4. Have active suicidal ideation with intent, based on Columbia-Suicide Severity Rating Scale (C-SSRS assessment (severity score >3) at the Screening visit, confirmed by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0 prior to randomization. Participants will be discharged if actively suicidal, and appropriate follow-up will be arranged.
5. Have made a medically significant suicide attempt (i.e., one that had a significant possibility of causing death or permanent harm in the absence of intervention) within the past 12 months, based on Screening C-SSRS assessment and confirmation by the Investigator. (Note: this criterion will be reassessed at each visit that occurs prior to Day 0, and on Day 0 prior to randomization. Participants will be discharged if actively suicidal, and appropriate follow-up will be arranged.)
6. Have a family history (first degree relatives) of schizophrenia, schizoaffective disorder, or bipolar disorder type 1.
7. Have a history of hallucinogen use disorder.
8. Have a history of hallucinogen persisting perceptual disorder (HPPD).
9. Have any use of classic psychedelics in the past 1 year.
10. Have > 25 lifetime uses of classic psychedelics.
11. Incarcerated or have pending legal action that could prevent participation in study activities.
12. Are court-mandated to complete residential treatment at SHH
13. Are unable or unwilling to discontinue taking any protocol-prohibited medications and supplements. (A detailed list of exclusionary medications is found in Section 6.5 of the protocol) Prohibited medications and supplements must have been stopped for at least 5 elimination half-lives or 14 days, whichever is longer, prior to Day 0 (Note: : Psychiatric medications will not be discontinued or changed in order to allow study participation. Concomitant medications will be reassessed on Day 0. Any patient who has started prohibited medications will be discharged from the study.)
14. Have a known allergy or hypersensitivity to psilocybin or any of the materials contained in the IP used in the study.
15. Have an allergy, hypersensitivity, or other contraindication that would preclude safe treatment of acute hypertension, anxiety, or psychotic symptoms if necessary during or immediately after the IP Administration Session, using the adjunctive medications used in this study to treat these symptoms (i.e., unable to take captopril and unable to take clonidine; unable to take diazepam and unable to take lorazepam; or unable to take olanzapine).
16. Have any other medical, psychiatric, or psychosocial disorder, symptom, condition, or situation that is likely to interfere with the establishment of rapport, adherence to study requirements, or safe administration of psilocybin or fMRI scanning, based on the judgement of the Investigator. (Note: This criterion will be reassessed on Day 0. Those not meeting the criterion will not be randomized but may be rescheduled once within 14 days if the criterion is likely to resolve within 14 days in the judgement of the Investigator.)
17. Inability to safely complete fMRI sessions (MRI screening form)
18. Any history of severe traumatic brain injury (assessed using the Ohio State University Traumatic Brain Injury (TBI) Identification [OSU TBI-ID] modified). (Note: If current (past 12 months) mild/moderate TBI and CSI score >/=12 (for either lifetime month or current month), the PI will determine eligibility.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in the alcohol cue-induced Blood-oxygen-level dependent (BOLD) signal in the lateral prefrontal cortex (PFC) | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the alcohol cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in the alcohol cue-induced BOLD signal change in the caudate | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the alcohol cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in alcohol cue-induced BOLD signal change in the ventromedial PFC (vmPFC) | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the alcohol cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in alcohol cue-induced BOLD signal change in the insula | Baseline, Day 2
  The blood-oxygen-level-dependent (BOLD) signal, detected in fMRI, reflects changes in deoxyhemoglobin driven by localized changes in brain blood flow and blood oxygenation, which are coupled to underlying neuronal activity by a process termed neurovascular coupling.
Percent change in negative affective cue-induced BOLD signal change in the dorsomedial PFC (dmPFC) | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the alcohol cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in negative affective cue-induced BOLD signal change in the supramarginal gyrus | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the negative affective cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in negative affective cue-induced BOLD signal change in the amygdala | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the negative affective cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in negative affective cue-induced BOLD signal change in the insula | Baseline, Day 2
  Percentage change in the BOLD signal is the difference in fMRI signal between the baseline condition (B) and the negative affective cue-induced task condition (T); percent signal change = (T-B)/B×100%. A positive value of the percentage change in BOLD signal indicates up-regulation of BOLD signal.
Percent change in alcohol cue-induced functional connectivity in prespecified regions of interest (ROI) | Baseline, Day 2
  ROI include the ventral striatum, lateral PFC (dlPFC and IFG), and caudate with target clusters in the PFC, ACC, and sensorimotor cortex (S1 and M1).
Percent change in negative affective cue-induced functional connectivity in prespecified regions of interest (ROI) | Baseline, Day 2
  ROI include the ventral striatal and amygdala with target clusters in temporal and occipital regions relative to placebo.
Percent change in the frequency of failed response inhibition | Baseline, Week 4
  A Go/NoGo task will be used as an objective measure of response inhibition. This task includes alcohol, non-alcohol, and neutral stimuli. The Go/No-go task requires participants to respond by pressing a button when they see a "go" signal, and not respond when they see the "no-go" signal. The key behaviour measured with this experiment is the participants' ability to withhold a response on No-go trials and the frequency of their failed responses.
Change in discounting rate (log(k)) | Baseline, Week 4
  The discounting rate is derived from the Delay Discounting Task. Delay discounting tasks provide a measure of the temporal window and examine the devaluation of awards as a function of the delay to the receipt. The task includes 80 items requiring a choice between a delayed reward of $100 and smaller immediate rewards (ranging from $10 to $99, at delays ranging from one to 365 days. Discounting rates will be measured and pre-post differences will be assessed. Higher k values indicate higher impulsive decision-making.
Change in number of set-shifting errors | Screening, Week 4
  Set-shifting errors are measured by the The Penn Conditional Exclusion Test (PCET). The PCET will be used as an objective measure of cognitive flexibility. A decrease in set-shifting errors equates to increased cognitive flexibility, while an increase in set-shifting errors equates to decreased cognitive flexibility.
Average number of no heavy drinking days | Week 24
  Outcome will be measured using the Timeline Followback (TLFB) interview-based assessment. The TLFB derives subjects' retrospective daily estimates of alcohol consumption patterns. Using a calendar as a visual aid, special events, and other memory cues, subjects are guided through the process of recalling and reporting daily drinking estimates.
Change in phosphatidyl ethanol (PEth) blood levels | Baseline, Week 12
Change in carbohydrate-deficient transferrin (CDT) blood levels | Baseline, Week 12
Change in the Drinker Inventory of Consequences questionnaire (DrInC-2R) total score | Baseline, Week 24
  DrInC-2R is a validated self-report questionnaire consisted of 50 questions to measure adverse consequences of alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal as well as frequency of these consequences (answers given on frequency scale grade from 0-3: 0 - never, 1 - once or a few times, 2 - once or twice a week 3 - daily or almost daily). Higher scores indicate greater levels of alcohol-related problems.
Change in PSQI global score | Baseline, Week 24
  Sleep quality is measured by the Pittsburgh Sleep Quality Index (PSQI) . The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The 19 items are grouped into 7 components, including (1) sleep duration, (2) sleep disturbance, (3) sleep latency, (4) daytime dysfunction due to sleepiness, (5) sleep efficiency, (6) overall sleep quality, and (7) sleep medication use. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction.
  Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep.
Change in patient's self-assessed quality of life (by the SF-36 Questionnaire) | Baseline, Week 24
  The Short Form Health Survey (SF-36) is a validated 36 item self-report Quality of Life Questionnaire that measures eight multi-item dimensions of health: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain, and general health perception. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Change in Alcohol craving score | Baseline, Week 24
  The alcohol cravings score will be assessed using the Penn Alcohol Craving Scale (PACS). The PACS consists of 5 questions with sub-scales ranging from 0 (never) to 6 (nearly all of the time). Scores greater than 20 were considered to meet diagnostic criteria for craving for a diagnosis of Substance Use Disorder.
Change in negative affect score | Baseline, Week 24
  Negative affect will be assessed using the negative affect scale of the Positive and Negative Affect Schedule (PANAS) which is a 10-item measure of negative emotions on a scale of 1 ("very slightly or not at all) to 5 ("extremely"). Total scores can range from 10 - 50, with higher scores representing higher levels of NA and reflect a dimension of general distress summarising a variety of negative states such as anger, guilt, or anxiety.
Change in impulsivity score (Barratt impulsivity scale by the subscales and by the total score) | Baseline, Week 24
  Impulsivity will be assessed using the Barratt impulsivity scale (BIS-11), a validated self-report questionnaire composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Items are scored on a 4-point scale: Rarely/Never = 1, Occasionally = 2, Often = 3, Almost Always/Always = 4. Total score is assessed. The total scores can range from 30 to 120. The higher total score corresponds to the more impulsive behavior

SECONDARY OUTCOMES:
Average number of no drinking days | Week 24
  Outcome will be measured using the Timeline Followback (TLFB) interview-based assessment. The TLFB derives subjects' retrospective daily estimates of alcohol consumption patterns. Using a calendar as a visual aid, special events, and other memory cues, subjects are guided through the process of recalling and reporting daily drinking estimates.
Percentage of heavy drinking days | Week 24
  Outcome will be measured using the Timeline Followback (TLFB) interview-based assessment. The TLFB derives subjects' retrospective daily estimates of alcohol consumption patterns. Using a calendar as a visual aid, special events, and other memory cues, subjects are guided through the process of recalling and reporting daily drinking estimates.
Average number of drinks per day | Week 24
  Outcome will be measured using the Timeline Followback (TLFB) interview-based assessment. The TLFB derives subjects' retrospective daily estimates of alcohol consumption patterns. Using a calendar as a visual aid, special events, and other memory cues, subjects are guided through the process of recalling and reporting daily drinking estimates.
Percentage of abstinent days | Week 24
  Outcome will be measured using the Timeline Followback (TLFB) interview-based assessment. The TLFB derives subjects' retrospective daily estimates of alcohol consumption patterns. Using a calendar as a visual aid, special events, and other memory cues, subjects are guided through the process of recalling and reporting daily drinking estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bogenschutz, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Silver Hill Hospital, New Canaan, Connecticut
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon request and approval by the NIH Data Access Committee immediately following article publication or as required by a condition of awards and agreements supporting the research. The NIH will provide access to scientific investigators for research purposes. Investigators requesting shared data must be affiliated with an NIH-recognized research institution (in the NIH's eRA Commons) that maintains an active FWA, and complete and submit a Data Use Certification approved by an authorized institutional business official with signature authority. Once approved, researchers will be granted access to the entire collection of shared data in the NDA research clusters requested. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Investigators requesting shared data must be affiliated with an NIH-recognized research institution (in the NIH's eRA Commons) that maintains an active FWA, and complete and submit a Data Use Certification approved by an authorized institutional business official with signature authority. This request will then be reviewed by the Data Access Committee (DAC). Once approved, researchers will be granted access to the entire collection of shared data in the NDA research clusters requested.
URL: https://nda.nih.gov/